CLINICAL TRIAL: NCT02764502
Title: Identification of Epidural Space Description of New Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osama Ali Ibraheim (Other)
Responsible Party: Sponsor-Investigator, Osama Ali Ibraheim, Professor Of Anesthesia, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 010007
Record Dates: First submitted 2016-04-10; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Anesthesia
Keywords: Epidural Identification pressure gauge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pressure Gauge Manometer (Experimental): Tuohy needle is introduced into intervertebral space at the level of L3-L4 up to the interspinous ligaments . The needle is advanced slowly using both hands while monitoring the manometer reading and is stopped when the pressure suddenly dropped ( the pressure usually drops by 5-10 mm Hg when the tip of the needle inters the epidural space ).
  Interventions: Device: Pressure Gauge Manometer

INTERVENTIONS:
Device: Pressure Gauge Manometer — Identification of epidural space

SUMMARY:
Introduction Several attempts have been made to improve or facilitate epidural space detection beside conventional loss of resistant technique. Recently many sophisticated equipment's and techniques have been described which did not received widespread popularity.

Objectives The Investigator describes and assesses the validity of using Pressure Gauge Manometer to confirm correct detection of lumber epidural space, in an inexpensive way.

Methods Tuohy needle is introduced into intervertebral space at the level of L3-L4 up to the interspinous ligaments ( nearly 2cm mark on the needle).A3-way stopcock is connected to the hub of Tuohy needle with the in-line port of the stopcock attached to an air-filled 10 ml syringe. Using a 75 cm extension tube set and create a 30 mm Hg pressure gradient between manometer and the tip of epidural needle , the needle is advanced slowly using both hands while monitoring the manometer reading and is stopped when the pressure suddenly dropped ( the pressure usually drops by 5-10 mm Hg when the tip of the needle inters the epidural space ).

DETAILED DESCRIPTION:
• A total of 60 consecutive ASA class 1& II patients of ages between 28-68 years scheduled for elective surgery under lumber epidural anesthesia or under general anesthesia with planned post-operative epidural analgesia were enrolled in this study.

Patients with known coagulation disorder, allergy to local anesthetics, skin lesions at the puncture side, or neuromuscular disease were not included.

Patients are placed in sitting position and American society of anesthesiologists standard monitors attached. After skin preparation, draping, and local anesthetic infiltration, an epidural Tuohy needle is introduced into intervertebral space at the level of L3-L4 up to the interspinous ligaments ( nearly 2cm mark on the needle). Fig 1 A3-way stopcock is connected to the hub of Tuohy needle with the in-line port of the stopcock attached to an air-filled 10 ml syringe. Using a 75 cm extension tube set the side port is connected to the Pressure Gauge Manometer held by the assistant. The stopcock is turned so that the needle is in direct continuity with both syringe and pressure Gage manometer. The syringe is used to create a 30 mm Hg pressure reading on the manometer, the stopcock then is turned into "open" to manometer and Tuohy needle and "close" to syringe.

With this 30 mm Hg pressure gradient between manometer and the tip of epidural needle, the needle is advanced slowly using both hands while monitoring the manometer reading and is stopped when the pressure changes ( the pressure usually drops by 5-10 mm Hg when the tip of the needle inters the epidural space ).

The 3-way is then removed and local anesthetic is injected for single shot epidural block or catheter is introduced in the conventional manner and secured by adhesive tap.

Procedure was performed by anesthetists of different levels of experience (consultant, specialist, resident).

Demographic data and type of surgery is recorded along with time of the technique, number of passes required to enter the epidural space, any false LOR, insertion difficulties, accidental dural puncture, or any other complication occurred.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1& II patients of ages between 28-68 years scheduled for elective surgery under lumber epidural anesthesia or under general anesthesia with planned post-operative epidural analgesia were enrolled in this study.

Exclusion Criteria:

* Patients with known coagulation disorder, allergy to local anesthetics, skin lesions at the puncture side, or neuromuscular disease were not included

Ages: 28 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Success of the technique. | 10 minutes after the technique.
  For epidural catheter placement success of the technique is defined as the installation of sensory block after the end of surgery.

SECONDARY OUTCOMES:
The physician satisfaction with the technique (Definitely not, Not completely, Yes) | 12hours after the end of the technique

CONTACTS AND LOCATIONS:
Overall Officials: Osama A Ibraheim, MD, Principal Investigator — Assiut University College of medicine
Locations (1):
- Assiut University ,Faculty Of Medicine ,Anesthesia Department, Egypt, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes